CLINICAL TRIAL: NCT00441506
Title: Effects of Daily Interruption of Sedatives in Critically Ill Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PP04
Record Dates: First submitted 2007-02-28; First posted 2007-03-01 (Estimated); Last update posted 2010-08-24 (Estimated); Status verified 2007-02

CONDITIONS: Critical Illness
Keywords: interruption; critically ill; sedation; pediatrics; critically ill, ventilated children
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: daily interruption of sedatives

SUMMARY:
Critically ill children are often sedated in order to relieve them from anxiety and discomfort, and to facilitate their care. There is little information on the effects of prolonged and continuous use of sedatives and analgesic agents in critically ill children. In adult intensive care unit (ICU) patients, daily interruption of sedative infusions accelerates recovery resulting in a reduction in the average duration of mechanical ventilation of 2.4 days as well as a reduction in average ICU length of stay of 3.5 days. These results were achieved without an increased rate of adverse events potentially linked to less sedation and associated with a reduction of common complications of critical illness and without negative psychological effects.

It is unknown whether these results can be extrapolated to critically ill children. Moreover, the possible risk of complications associated with less sedation, such as accidental self-extubation, is probably higher in children. Also, the need for intermittent bolus administrations in children treated with intermittent sedation could nullify the reduction in the use of sedatives.

It is unknown if daily interruption of sedatives is feasible in critically ill children. The researchers studied the effects of daily interruption of sedatives in critically ill children on the total amount of sedatives used and risks of complications.

ELIGIBILITY:
Inclusion Criteria:

* Intubated and mechanically ventilated for > 24 hours
* Expect further mechanical ventilation for > 48 hours
* Receiving midazolam and morphine for sedation
* Written informed consent given by parents

Exclusion Criteria:

* Inclusion in another trial
* Transfer from an outside institution where sedatives had been administered
* Neuromuscular blockers
* Metabolic disease
* Neuromuscular disease
* Encephalopathy
* Epilepsy
* Pulmonary hypertension
* Neurotrauma
* Raised intracranial pressure
* Life expectancy less than a month/infaust prognosis

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2004-11; Primary Completion 2006-06 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
amount of (near) incidents | Until extubation or 28 days
total amount of sedatives administered | Until extubation or 28 days
time to wake up (after sedation is stopped), comfort scale | Until extubation or 28 days
BIS monitoring | Until extubation or 28 days

SECONDARY OUTCOMES:
time on ventilator | Until extubation or 28 days
LOS on ICU | Until extubation or 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Peter Pickkers, MD, PhD, Study Director — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Center, Nijmegen, Gelderland, Netherlands